CLINICAL TRIAL: NCT05216861
Title: Evaluation of a Collaborative Intervention to Promote Early Employer Contact and Return to Work Among People With Common Mental Disorders or Long-term Pain
Brief Title: Evaluation of a Collaborative Intervention to Promote Employer Contact and RTW Among People With CMD or Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Therese Hellman, PhD, Associate professor, Uppsala University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RFR-968570
Record Dates: First submitted 2022-01-17; First posted 2022-02-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pain, Chronic; Mental Disorder
MeSH Terms: conditions — Chronic Pain; Mental Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The rehabilitation coordinators are trained in the intervention (0,5 day).
  Interventions: Other: Demand and ability protocol
- Active comparator (Other): Participants in the experimental arm will be matched with controls from the Micro Data for the Analysis of Social Insurance register (MiDAS) from the Social Insurance Agency, Sweden.
  Interventions: Other: Collaborative interventions as usual

INTERVENTIONS:
Other: Demand and ability protocol — The intervention consists of a structured conversation between the patient and his immediate manager under the guidance of licensed medical staff (in this case REKO) with knowledge of the requirements of the patient's work and his/her current functional ability. The intervention takes about 90 minutes excluding preparation time for REKO.
  DAP consider the following domains; 1) mental and cognitive ability, 2) basic skills and social ability, 3) tolerance for physical conditions, 4) ability to work dynamically, 5) ability to work statically and 6) to be able to work certain times.
  Based on the above domains, a structured review is made of the balance between requirements and function in current work in order to identify possible adaptations and measures at the workplace. During the intervention, the work requirements and the patient's function/ability are identified on a three-point scale and in domains where there is thus an imbalance adjustments or changed tasks are identified.
  Arms: Experimental
Other: Collaborative interventions as usual — The rehabilitation coordinator conduct collaborative interventions as usual with patient and employer. This might be through phone calls are unstructured meetings.
  Arms: Active comparator

SUMMARY:
The overall aim of this cluster ranomized controlled trial is to investigate whether an intervention for collaboration between patient with CMD or chronic pain and employer (the Demand and Ability Protocol) can contribute to reduced sick leave and to increased health, work ability and trust in the managers. The intervention is delivered by rehabiliation coordinators at primary health care centres.

DETAILED DESCRIPTION:
The overall aim of this cluster ranomized controlled trial is to investigate whether an intervention for collaboration between patient with CMD or chronic pain and employer (the Demand and Ability Protocol) can contribute to reduced sick leave and to increased health, work ability and trust in the managers. The intervention is delivered by rehabilitation coordinators at primary health care centres.

Furthermore, the aim is to identify hindering and facilitating factors for feasibility, usability and implementation of the Demand and Ability Protocol intervention (DAP) in primary health care.

Research questions:

1. What is the effect of DAP for patients regarding sick leave, health, work ability, and trust in the manager compared to matched controls who do not recieve DAP?
2. How do patients and managers experience their participation in the intervention and how do they experience the usability of the DAP?
3. What facilitating and hindering factors exist for the introduction and implementation of DAP in primary health care, and how do rehabilitation coordinators (REKO) and medical doctors experience the feasibility and usability of the intervention?

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of CMD and/or chronic pain
* have a job
* be on full-time or part time sick leave
* accept the manager's involvement.

Exclusion Criteria:

* been on full-time sick leave for more than 6 months before the first contact with REKO

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Sick leave | From baseline until 12 months
  The total number of days on sick leave due to CMDs or chronic pain during the 12 month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Therese Hellman, PhD, Principal Investigator — Uppsala University
Locations (1):
- Region Uppsala, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No